CLINICAL TRIAL: NCT03110939
Title: A Phase III, Single Center Randomized Controlled Trial of Thoracic Surgery Combined With Intrathoracic Hyperthermic Perfusion for Advanced Lung Cancer / Esophageal Cancer
Brief Title: Thoracic Surgery Combined With Intrathoracic Hyperthermic Perfusion for Advanced Lung Cancer / Esophageal Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The principal investigator Dr.YinLi is working in other Hospital
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Yin Li, vice president of Henan Cancer Hospitan and director of thoracic surgery department, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HenanCH2016ct082
Record Dates: First submitted 2017-03-28; First posted 2017-04-12 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Esophageal Cancer; Lung Cancer; Hyperthermic Perfusion
MeSH Terms: conditions — Esophageal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hyperthermic perfusion group (Experimental): hyperthermic perfusion 1800-2000ml, normal saline, 45-48℃, 1 hour, speed 300-600ml/min (after standard surgery of advanced lung cancer/esophageal cancer)
  Interventions: Other: hyperthermic perfusion
- control group (No Intervention): standard surgery of advanced lung cancer/esophageal cancer

INTERVENTIONS:
Other: hyperthermic perfusion — hyperthermic perfusion 1800-2000ml, normal saline, 45-48℃, 1 hour, speed 300-600ml/min (after surgery of advanced lung cancer/esophageal cancer)
  Arms: hyperthermic perfusion group

SUMMARY:
The goal of this clinical research study is to explore whether intrathoracic hyperthermic perfusion after radical surgery could reduce local recurrence rate(13%) for advanced lung cancer / esophageal cancer. The safety of intrathoracic hyperthermic perfusion right after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must not have received any prior anticancer therapy of cancer.
2. expected R0 resection.
3. Histologic diagnosis of squamous cell thoracic esophageal carcinoma of T3-4, any N and any T, N1. (8th Union for International Cancer Control, Union for International Cancer Control(UICC)-TNM). Histologic diagnosis of non small cell lung cancer, T2-T3, any N. (8th Union for International Cancer Control, UICC-TNM)
4. Age ranges from 18 to 80 years.
5. Without operative contraindication.
6. Eastern Cooperative Oncology Group (ECOG) 0～2.
7. Signed informed consent document on file.

Exclusion Criteria:

1. Multiple primary cancer.
2. The subject cannot understand and sign the informed consent form(ICF).
3. Patients with concomitant hemorrhagic disease.
4. Any un expected reason for patients can't get operation.
5. Pregnant or breast feeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2019-04-05 (Estimated); Study Completion 2021-04-05 (Estimated)

PRIMARY OUTCOMES:
local recurrent rate | 3 years after surgery
  recurrent within thoracic cavity

SECONDARY OUTCOMES:
Total complication rate | 6 months after surgery
  The total complications mean anastomotic fistula, hydrothorax, pneumonia, pleural hemorrhage and cardiac together.
The Clavien-Dindo classification | 6 months after surgery
  the classification surgical complications after surgery/intrathoracic hyperthermic perfusion
mortality rate during operation/intrathoracic hyperthermic perfusion | during operation/intrathoracic hyperthermic perfusion
  mortality rate during operation/intrathoracic hyperthermic perfusion
vital signs during treatment | during operation/intrathoracic hyperthermic perfusion
  The heart rate, blood pressure and body temperature will be recorded every 10 mins during intrathoracic hyperthermic perfusion
mortality rate after treatment | 2 months after surgery/intrathoracic hyperthermic perfusion
  mortality rate after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided